CLINICAL TRIAL: NCT02915601
Title: Bicarbonate Administration in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1572
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Disease; Metabolic Acidosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Bicarbonate (Experimental): Participants assigned to oral sodium bicarbonate will receive 0.5 mEq/kg-lean body weight (LBW)/day for the entire 12 months. Participants will take ½ the daily dose in the morning and the other ½ in the evening. The number of capsules will be rounded to the nearest whole capsule. To reduce pill burden and increase compliance the maximum number of pills per day will be six.
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): Subjects randomly assigned to placebo will take the same number of capsules as if they were assigned to receive 0.5 mEq/kg-LBW/day of sodium bicarbonate. Participants will take ½ the daily dose in the morning and the other ½ in the evening. The number of capsules will be rounded to the nearest whole capsule. To reduce pill burden and increase compliance the maximum number of pills per day will be six.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate
  Arms: Sodium Bicarbonate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Low serum bicarbonate levels, even within the normal laboratory range, are strongly associated with increased risks of hypertension, endothelial dysfunction, cardiovascular disease and death. The current proposal will investigate whether bicarbonate administration in patients with chronic kidney disease (CKD) will improve the health and function of arteries and reduce the size of the left ventricle of the heart. Overall, the proposed research will provide important new scientific evidence upon which physicians can base recommendations to patients with CKD to decrease the risk of developing cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Serum bicarbonate 22-25 mEq/L on 2 separate measurements (at least 1 day apart)
* CKD stage 3B or 4 at time of screening (eGFR 15-44 ml/min/1.73m2)
* Blood pressure <130/80 mm Hg prior to randomization
* BMI < 40 kg/m2 (FMD measurements can be inaccurate in severely obese patients).
* Able to provide consent
* Stable anti-hypertensive regimen for at least one month prior to randomization
* Not taking medications that interact with agents administered during experimental sessions (e.g. sildenafil interacts with nitroglycerin).

Exclusion Criteria:

* Use of chronic daily oral alkali within the last 3 months (including sodium bicarbonate, calcium carbonate or baking soda)
* Uncontrolled hypertension
* Serum potassium < 3.3 or ≥ 5.5 mEq/L at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known EF ≤30%, or hospital admission for heart failure within the past 3 months
* Factors judged to limit adherence to interventions
* Anticipated initiation of dialysis or kidney transplantation within 12 months
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Chronic use of supplemental oxygen
* Use of immunosuppression in past 3 months
* Metal implant or implanted electrical device (patient will be unable to get MRI)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.

REFERENCES:
- [Derived] Zhang A, Furgeson S, Shapiro A, Bjornstad P, You Z, Tommerdahl KL, Dixon A, Stenson E, Oh E, Kendrick J. Assessing Cognition in CKD Using the National Institutes of Health Toolbox. Kidney360. 2024 Jun 1;5(6):834-840. doi: 10.34067/KID.0000000000000440. Epub 2024 Apr 3. PMID 38568010
- [Derived] Perez L, You Z, Kendrick J. Association of Plant-Based Protein Intake with Cognitive Function in Adults with CKD. Kidney360. 2023 Nov 1;4(11):1554-1561. doi: 10.34067/KID.0000000000000278. Epub 2023 Oct 27. PMID 37889573
- [Derived] Kendrick J, You Z, Andrews E, Farmer-Bailey H, Moreau K, Chonchol M, Steele C, Wang W, Nowak KL, Patel N. Sodium Bicarbonate Treatment and Vascular Function in CKD: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2023 Aug 1;34(8):1433-1444. doi: 10.1681/ASN.0000000000000161. Epub 2023 May 25. PMID 37228030

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Bicarbonate: Participants assigned to oral sodium bicarbonate will receive 0.5 mEq/kg-lean body weight (LBW)/day for the entire 12 months. Participants will take ½ the daily dose in the morning and the other ½ in the evening. The number of capsules will be rounded to the nearest whole capsule. To reduce pill burden and increase compliance the maximum number of pills per day will be six.
  Sodium bicarbonate
- Placebo: Subjects randomly assigned to placebo will take the same number of capsules as if they were assigned to receive 0.5 mEq/kg-LBW/day of sodium bicarbonate. Participants will take ½ the daily dose in the morning and the other ½ in the evening. The number of capsules will be rounded to the nearest whole capsule. To reduce pill burden and increase compliance the maximum number of pills per day will be six.
  Placebo
Period: Overall Study
Arm/Group | Sodium Bicarbonate | Placebo
Started | 55 | 54
Completed | 44 | 46
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.5) | 62.6 (10.7) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 42 | 44 | 86
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Artery Flow Mediated Dilation
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 44 | 46
percentage
  Baseline | 3.99 (4.8) | 3.78 (4.3)
  12 months | 4.25 (3.51) | 4.43 (3.9)

2. Primary Outcome: Change in Aortic Pulse Wave Velocity
Time Frame: Measured at baseline,12 months
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 44 | 46
cm/sec
  Baseline | 998.3 (447.5) | 994.8 (373.5)
  12 months | 1067.2 (457.9) | 983.4 (347.7)

3. Secondary Outcome: Change in Left Ventricular Mass Index
Time Frame: Measured at baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: g/m2
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 44 | 46
g/m2
  Baseline | 57.4 [51.5 to 67.9] | 59.4 [51.4 to 76.1]
  12 months | 57.2 [53.1 to 66.8] | 67.6 [51.6 to 78.3]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Sodium Bicarbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 1/54
Serious Adverse Events (participants affected / at risk) | 7/55 | 7/54
Other Adverse Events (participants affected / at risk) | 36/55 | 28/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate (N=55) | Placebo (N=54)
Hospitalizations (Infections and infestations) | 1 (1) | 1 (1)
Hospitalizations (Cardiac disorders) | 1 (1) | 2 (2) — Volume overload MI/stroke
Hospitalization (Gastrointestinal disorders) | 1 (1) | 2 (2) — Planned surgery Ileus
Hospitalization (Renal and urinary disorders) | 0 (0) | 1 (1) — acute on chronic renal failure
Hospitalization (Endocrine disorders) | 2 (2) | 0 (0) — High/low glucose levels
Hospitalization (Vascular disorders) | 1 (1) | 0 (0) — Loss of consciousness
Initiation of dialysis (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate (N=55) | Placebo (N=54)
Increase in diuretic therapy (Cardiac disorders) | 8 (8) | 7 (7)
Increase in antihypertensive therapy (Cardiac disorders) | 11 (11) | 12 (12)
High serum bicarbonate level >28 mEq/L (Renal and urinary disorders) | 13 (13) | 1 (1)
Low serum bicarbonate level < 20 mEq/L (Renal and urinary disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02915601/Prot_SAP_000.pdf